CLINICAL TRIAL: NCT01719523
Title: Open-Trial of EPI-743 for Adults With Tourette Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Rembrandt Foundation (Unknown); Edison Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120100953972412
Record Dates: First submitted 2012-10-29; First posted 2012-11-01 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Tourette Syndrome
Keywords: Tourette syndrome; Tics; Tic Disorders
MeSH Terms: conditions — Tourette Syndrome; Tics; Tic Disorders | interventions — alpha-tocotrienol quinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EPI-743 (Experimental): EPI-743- Participants will receive 200mg three times a day of EPI-743 for 2 weeks and then receive 300mg of EPI-743 for an additional 2 weeks.
  Interventions: Drug: EPI-743

INTERVENTIONS:
Drug: EPI-743

SUMMARY:
The purpose of this study is to examine the effects of EPI-743 on tic severity in adults with Tourette syndrome.

DETAILED DESCRIPTION:
Tourette syndrome (TS) is a childhood-onset neuropsychiatric disorder characterized by multiple motor and vocal tics that last for at least a year in duration. Currently, there exist several effective pharmacological treatments for childhood tics including alpha-2 agonist medications (guanfacine and clonidine) and neuroleptics (antipsychotic) medications. These medications, however, have significant side-effects and are only partially effective in treating tics.

EPI-743 is an orally absorbed small molecule that readily crosses into the central nervous system. It works by targeting an enzyme NADPH quinone oxidoreductase 1 (NQO1). Its mode of action is to synchronize energy generation in mitochondria with the need to counter cellular redox stress. EPI-743 has recently received orphan drug status from the U.S. Food and Drug Administration (FDA). The FDA has allowed an Expanded Access program to provide EPI-743 to seriously ill patients diagnosed with inherited respiratory chain diseases of the mitochondria.

The rationale for the use of this agent is indirect. Over the past 10 years, defects in mitochondrial oxidative phosphorylation (OXPHOS) have been implicated in a wide variety of neurodegenerative and neuromuscular diseases. One neurological symptom that has definitely been associated with OXPHOS is the movement disorder dystonia. A specific missense mutation in the mtDNA complex I (NADH dehydrogenase) gene, MTND6, has been linked to maternally inherited dystonia along with the companion phenotype, Leber's hereditary optic neuropathy. In addition, other mitochondrial diseases are also associated with movement disorders including Friedreich's ataxia (ataxia) and Leigh's disease (loss of head control and other motor skills). EPI-743 has been effective in treating children and adults with these diseases. Over time, many TS patients develop complex motor tics, which are sudden, more purposive appearing, stereotyped movements of variable duration. Examples are myriad and include facial gestures and movements such as brushing hair back, possibly in combination with head jerk, and body shrugs. Gyrating, bending, and twisting movements of the head or torso are also seen. These slow twisting movements are usually referred to as dystonic tics.

A second line of evidence concerns the potential therapeutic value N-acetyl-cysteine (NAC) in the treatment of neuropsychiatric conditions closely related to TS including Trichotillomania (TTM) and Obsessive-compulsive disorder [OCD]. Recent double-blind, placebo-controlled studies of NAC have provided evidence of efficacy in reducing the symptoms of trichotillomania (TTM) in adults [49]. The effect size in this 12-week study was strikingly large (d = 1.3). Trichotillomania, like TS, is considered to be an obsessive-compulsive spectrum disorder. Individuals with TTM experience urges prior to hairpulling, similar to the urges in TS. Case reports have also suggested the potential efficacy of NAC in treating OCD. NAC is hypothesized to have two possible mechanisms of action. NAC is converted to cystine, a substrate for the glutamate/cystine antiporter located on glial cells. The uptake of cystine by glia causes the release of glutamate into the extrasynaptic space, where it stimulates inhibitory metabotropic glutamate receptors on glutamatergic nerve terminals and thereby reduces the synaptic release of glutamate. NAC is also a precursor of glutathione, the major antioxidant in the brain. Through this mechanism NAC is hypothesized to improve OXPHOS. One effect of EPI-743's activity on NQO1 is restoration of cellular glutathione stores.

A third line of indirect evidence is that in postmortem brain studies, the two classes of interneurons that are reduced in number in the basal ganglia are "high energy" consuming cells, i.e., GABAergic, fast spiking internerons and cholinergic tonically active interneurons. Given the high energy demand associated with these cells perhaps their loss is partially due to defects in OXPHOS.

A fourth line of indirect evidence is that when EPI-743 is effective in treating mitochrondrial disease, brain regions with very low HMPAO uptake show a marked increase in uptake. In the case of TS (50 cases and 20 controls) HMPAO uptake was found to be reduced in the left caudate, anterior cingulate cortex and the left dorsolateral prefrontal cortex. Severity of tics was related to hypoperfusion of the left caudate and cingulate and a left medial temporal region.

ELIGIBILITY:
Inclusion Criteria:

* Adult between 18-65 years of age
* Meet DSM IV criteria for the diagnosis of Tourette's syndrome
* Significant current tic symptoms: YGTSS total tic score greater than or equal to 22 at baseline
* On stable psychiatric medication regimen for a minimum of 4 weeks prior to beginning the trial.
* Accepted method of birth control
* Willingness to participate in an HMPAO SPECT scan at baseline and after 4 weeks of treatment.

Exclusion Criteria:

* Comorbid bipolar disorder, psychotic disorder, substance use disorder, developmental disorder or intellectual disability (IQ<70).
* Recent change (less than 4 weeks) in medications that have potential effects on tic severity. Medication change is defined to include dose changes or medication discontinuation.
* Recent change in behavioral treatment for Tourette syndrome or comorbid conditions (i.e. OCD) within the last 4 weeks or initiation of behavioral therapy for tics within the last 12 weeks.
* Known hypersensitivity or previous anaphylactoid reaction to EPI-743 or any components in its preparation
* Positive pregnancy test or drug screening test
* Clinical history of bleeding disorder or abnormal baseline PT/PTT
* Hepatic insufficiency with LFTs greater than two times upper limit of normal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Yale Global Tic Severity Scale | Baseline
Yale Global Tic Severity Scale | 2 weeks
Yale Global Tic Severity Scale | 4 weeks

SECONDARY OUTCOMES:
Premonitory Urge for Tics Scale | Baseline
Yale-Brown Obsessive Compulsive Scale | Baseline
Connors Adult Attention Deficit Hyperactivity Rating Scale | Baseline
Hamilton Rating Scales for Depression and Anxiety | Baseline
Clinical Global Improvement | Week 4
Columbia Suicide Severity Rating Scale | Baseline
Adverse Events Rating Scale | Week 2
Premonitory Urge for Tics Scale | Week 2
Premonitory Urge for Tics Scale | Week 4
Adverse Events Rating Scale | Week 4
Yale-Brown Obsessive Compulsive Scale | Week 2
Yale-Brown Obsessive Compulsive Scale | Week 4
Connors Adult Attention Deficit Hyperactivity Rating Scale | Week 2
Connors Adult Attention Deficit Hyperactivity Rating Scale | Week 4
Hamilton Rating Scales for Depression and Anxiety | Week 2
Hamilton Rating Scales for Depression and Anxiety | Week 4
Clinical Global Improvement | Week 2
Columbia Suicide Severity Rating Scale | Week 2
Columbia Suicide Severity Rating Scale | Week 4

OTHER OUTCOMES:
HMPAO Uptake in Frontal-Striatal Circuit on SPECT Scan | Baseline
HMPAO Uptake in Frontal-Striatal Circuit on SPECT Scan | Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Bloch, MD, MS, Principal Investigator — Yale University
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States